CLINICAL TRIAL: NCT01557595
Title: Evening Use of Polarized Glasses Designed to Filter Out Blue Light in Attention Deficit Hyperactivity Disorder - Delayed Circadian Rhythm Disorder Patients
Brief Title: Blue Wavelength Light-blocking Glasses in ADHD-Insomnia
Acronym: ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Rachel Fargason, MD, MD, Associate Professor Psychiatry, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X110825016
Record Dates: First submitted 2012-02-16; First posted 2012-03-19 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Attention Deficit Hyperactivity Disorder; Delayed Sleep Phase Type Circadian Rhythm Sleep Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adults with ADHD (Experimental): Participants will be given polarized glasses (yellow "sun"- glasses) which filter out blue light to wear only from sundown until bedtime for two weeks. Subjects will 19 years or older and have ADHD
  Interventions: Device: Polarized glasses designed to filter out blue light

INTERVENTIONS:
Device: Polarized glasses designed to filter out blue light — Participants will be given polarized glasses (yellow "sun"- glasses) which filter out blue light to wear only from sundown until bedtime for two weeks. They will be instructed to turn off fluorescent lights and only use household lamps for evening activities. They will be instructed not to drive while wearing the glasses. In addition to the oral instructions, they will also be given a written "Instruction Sheet." Any oral insomnia agent will be held throughout the study, otherwise they are to follow their usual evening routines. This is an alternative treatment already in use in Dr. Fargason's practice for those patients who don't want to take sleep medications. This research focuses on the effectiveness of this treatment and involves questionnaires to do so.
  Other Names: Lowbluelights.com eyewear

SUMMARY:
Patients with ADHD often report staying up late on the computer, watching TV, or using other electronic devices, all strong emitters of blue light which may be contributing to the delayed sleep onset times seen in some of these patients. Evening use of polarizing glasses which filter out blue light may decrease the contribution of environmental light late at night to delayed bedtime. This is a treatment that Dr. Fargason uses when patients do not want to use sleep medication to help them fall asleep. The purpose of this study is to evaluate the effectiveness of this treatment by use of sleep diaries and sleep questionnaires.

DETAILED DESCRIPTION:
Blue light in the 460-480 nm range is known to suppress melatonin onset and signal alerting mechanisms in the brain. Patients with ADHD often report staying up late on the computer, watching TV, or using other electronic devices, all strong emitters of blue light which may be contributing to the delayed sleep onset times seen in these patients. (Ramelteon for insomnia due to ADHD, R Fargason, K Gamble, K Avis, R Besing, R May, Psychopharmacology Bulletin, submitted March 2011). Dr. Fargason is using polarized glasses to treat patients who do not want to take sleep medications to facilitate earlier sleep onset.

At the screen visit, following the informed consent procedure, ADHD + Delayed CRSD participants will fill out the demographic sheet and will be interviewed by the investigator regarding their history of sleep medications. If they are currently taking sleep medications and wish to stop taking them in order to participate in the study, they will be instructed how to safely do this. Following a two week washout period, participants will be given 7 wake up and bedtime diaries to complete. If the participant has not been on sleep medications for the last two weeks, they will receive the 7 sets of diaries at the screen visit and instructed to complete them twice daily.

At the baseline visit, the diaries will be retrieved. The participants will complete a baseline Pittsburgh Sleep Quality Index (PSQI), and will be given 14 sets of wake up and bedtime diaries. Participants will also be given polarized glasses which filter out blue light to wear only from sundown until bedtime for two weeks. They will be instructed to turn off fluorescent lights and only use household lamps for evening activities. They will be instructed not to drive while wearing the glasses. In addition to the oral instructions, they will also be given a written "Instruction Sheet." Any oral insomnia agent will be held throughout the study, otherwise they are to follow their usual evening routines. This is an alternative treatment already in use in Dr. Fargason's practice for those patients who don't want to take sleep medications. This research focuses on the effectiveness of this treatment and involves questionnaires to do so.

The diaries will then be filled out daily for 2 weeks; days with extenuating circumstances (i.e. nighttime trip to ER) will be noted; the PSQI will be filled out again at the 2 week termination visit. All forms will be collected with the glasses at the 2 week visit. This data is being gathered in patients who have remained in clinical treatment with Dr. Fargason and view this as an opportunity to have a free trial of the polarizing glasses before purchasing them for their own use to advance their sleep phase. This idea was prompted by the patients' eagerness to try the glasses clinically and hence avoid need for sleep medication.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age and older
* Diagnosis of ADHD and DCRD
* Willingness to sign consent and participate in the study

Exclusion Criteria:

* No sleep medication for previous two weeks before screen visit (Can enroll if willing to undergo washout period)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Fargason, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Adults With ADHD: Participants age 19 and older with a diagnosis of ADHD, in a generally healthy medical condition were recruited. Daily bedtime, wake-up time, and compliance diaries were used to assess sleep quality and timing during a baseline observation week and a 2-week intervention period. The Pittsburgh Sleep Quality Index (PSQI) was administered following baseline and intervention. The intervention protocol consisted of use of blue wavelength-blocking glasses and a moderate lighting environment during evening hours.
Period: Overall Study
Arm/Group | Adults With ADHD
Started | 22
Completed | 14
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Adults With ADHD
Number analyzed (Participants) | 22
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 22
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) was measured at the end of the baseline assessment week and again after the intervention. The PSQI is a validated self-rating instrument assessing aspects of sleep quality. The PSQI is considered appropriate in edentifying new onset insomnia in the clinical setting.
  units on a scale | 11.15 (3.50)

OUTCOME MEASURES:

1. Primary Outcome: Pittsburgh Sleep Quality Index (PSQI) at 2 Weeks After Baseline
Description: The PSQI is a validated self-rating instrument assessing aspects of sleep quality.Minimum score 0 (better); maximum score 21 (worse) < or = 5 associated with good sleep quality; > 5 associated with poor sleep quality. The PSQI is considered appropriate in identifying "new-onset" insomnia in the clinical setting.
Time Frame: 2 weeks post baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Adults With ADHD: Participants age 19 and older with a diagnosis of ADHD, in a generally healthy medical condition were recruited.
Arm/Group | Adults With ADHD
Number analyzed (Participants) | 14
units on a scale | 4.54 (3.15)

ADVERSE EVENTS:
Arm/Group | Adults With ADHD
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 2/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adults With ADHD (N=22)
intermittent headache (General disorders) | 1 — Mild intermittent headache, possibly related to intervention, non-serious, resolved by end of study participation.
pain on bridge of nose (General disorders) | 1 — Mild pain on surface of bridge of nose, related to intervention, resolved by end of study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes